CLINICAL TRIAL: NCT05613608
Title: Alcohol Use Disorder and Cannabis: Testing Novel Harm Reduction Strategies
Brief Title: Alcohol Use Disorder and Cannabidiol
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-1894; R01AA029606 (NIH)
Record Dates: First submitted 2022-10-28; First posted 2022-11-14 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Alcohol Use Disorder
Keywords: alcohol; cannabidiol; cbd; cannabis
MeSH Terms: conditions — Alcoholism; Color Vision Defects; Marijuana Abuse | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: This is a double-blind, placebo-controlled, parallel group study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Full-Spectrum Cannabidiol (Active Comparator): 210mg/day of full-spectrum cannabidiol, containing less than 0.3% THC.
  Interventions: Drug: Cannabidiol
- Broad-Spectrum Cannabidiol (Active Comparator): 210mg/day of full-spectrum cannabidiol, containing 0.0% THC.
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): 210mg/day of hemp seed oil with no cannabinoids present.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — The current study will directly test the hypothesis that a moderate dose of CBD leads to a reduction in alcohol consumption, alcohol craving, peripheral markers of inflammation, and anxiety.
  Arms: Broad-Spectrum Cannabidiol; Full-Spectrum Cannabidiol
Drug: Placebo — Placebo arm.
  Arms: Placebo

SUMMARY:
This is a double-blind, placebo-controlled, parallel group study designed to assess the efficacy of full spectrum CBD and broad spectrum CBD, compared to a placebo control (PC), to reduce drinking in participants with alcohol use disorder. If eligible for the study, subjects will be randomized to receive one of the conditions for 12 weeks.

DETAILED DESCRIPTION:
To better understand the effects of hemp-derived CBD with and without a small amount of THC, we propose a Phase II randomized clinical trial (RCT) to examine the safety, tolerability, and clinical effects of Full Spectrum CBD (fsCBD, contains less than 0.3% THC) vs. Broad Spectrum CBD (bsCBD, does not contain THC), vs. a matching placebo in a population of AUD subjects.

This is a double-blind, placebo-controlled, parallel group study designed to assess the efficacy of fsCBD and bsCBD, compared to a placebo control, to reduce drinking in participants with moderate alcohol use disorder according to the DSM-V. If eligible for the study, subjects will be randomized to receive one of the conditions for 12 weeks. The current study will test the hypothesis that a moderate dose of CBD leads to a reduction in alcohol consumption, alcohol craving, peripheral markers of inflammation, and anxiety. It is further hypothesized that CBD will lead to increased sleep duration and quality among individuals with AUD who want to quit or reduce their drinking. The study will also determine whether the small amount of THC found in full spectrum hemp-derived CBD products produces any negative effects.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥21 years old.
2. Meets Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-V) criteria for current Alcohol Use Disorder (AUD) of at least moderate severity (i.e., 4 or more DSM-V symptoms).
3. Expresses desire to reduce or quit drinking.
4. If male, reports drinking, on average, at least 15 standard alcoholic drinks per week prior to screening; if female, reports drinking, on average, at least 10 standard drinks per week prior to screening.
5. Able to attend in-person visits at the study site.
6. Participants reporting current nicotine use in any form will be included.

Exclusion Criteria:

1. Self-reported DSM-V diagnosis of any other substance use disorder.
2. Self-report illicit/recreational use of cocaine, methamphetamines, amphetamines, MDMA, opioids, or benzodiazepines in the last 30 days.
3. Daily cannabis use.
4. Uses CBD products for medical reasons.
5. Self-reports or indicates having a serious DSM-V psychiatric disorder, including panic disorder, obsessive/compulsive disorder, post-traumatic stress disorder, bipolar affective disorder, schizophrenia, cluster B personality disorders (borderline, antisocial, histrionic, narcissistic), eating disorders, or any other psychotic mental disorder.
6. Endorsing item 2 on the C-SSRS measure of suicide risk.
7. Currently taking any of the following medications:

   1. Those known to have a major interaction with Epidiolex.
   2. Acute treatment with any antiepileptic medications.
   3. Medication known to affect alcohol intake (e.g., disulfiram, naltrexone, acamprosate, and/or topiramate).
8. Self-reported history of severe alcohol withdrawal (e.g., seizure, delirium tremens).
9. Clinically significant medical problems in the last six months, such as cardiovascular, renal, gastrointestinal, or endocrine problems, that would impair participation or limit medication ingestion.
10. Current or past alcohol-related medical illness, such as gastrointestinal bleeding, pancreatitis, hepatocellular disease, or peptic ulcer.
11. Females of childbearing potential who are pregnant, nursing, or who are not using a reliable form of birth control.
12. Current charges pending for a violent crime (not including DUI-related offenses).
13. Lack of a stable living situation.
14. Lack of access to internet.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change in Drinks per Drinking Day | 0-12 weeks
  The Time Line Follow Back is a calendar-assisted measure that can be used to assess alcohol, tobacco, cannabis, and other substance use. The investigators will use this measure to create the Drinks per Drinking Day variable.
Change in Alcohol Use Disorder | 0-12 weeks
  The AUDIT consists of ten questions that cover such domains as alcohol consumption, drinking behavior, adverse psychological reactions, and alcohol-related problems.
Change in Alcohol Craving | 0-12 Weeks
  The Penn Alcohol Craving Scale (PACS) will be used to assess changes in alcohol craving.

SECONDARY OUTCOMES:
Change in Cue-reactivity | 0-12 weeks
  Cue-elicited urge to drink will be assessed using the cue-reactivity assessment, per protocol (Hutchison, 2006).
Change in Anxiety | 0-12 weeks
  The Depression Anxiety Stress Scale is a 21-item self-report instrument for measuring the three related negative emotional states of depression, anxiety, and tension/stress. Participants rate their anxiety on a scale from 1 (Did not apply to me at all) to 4 (Applied to me very much/most of the time), with higher scores indicating worse outcomes.
Change in Pain Levels | 0-12 weeks
  The PROMIS Numeric Rating Scale v1.0 - Pain Intensity - 1a consists of a single item rating pain on average over the past 7 days from 0 (no pain) to 10 (worst pain you can think of). Participants are also asked to rate the impact of their pain in the last 7 days. The PROMIS Short Form v1.1 - Pain Interference - 6b rates pain on a scale from 1 (not at all) to 5 (very much), as it refers to the degree to which pain limits or interferes with subjects' physical, mental, and social activities.
Change in Sleep Disturbance | 0-12 weeks
  The PROMIS Short Form v.1.0 - Sleep Disturbance - 4a will be used to measure self-reported perceptions of sleep quality, depth, and restoration within the past seven days. This includes perceived difficulties falling asleep and staying asleep, as well as sleep satisfaction.
Change in Impaired Control Scale (ICS) | 0-12 Weeks
  The Impaired Control Scale will assess impulsivity, awareness of compulsion to drink, and control over drinking behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Kent Hutchison, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be made available on the NIMH Data Archive.
Supporting Information: Analytic Code
Time Frame: The data will be submitted twice yearly with the first submission to occur in April 2023. The data will be available on the NIMH Data Archive indefinitely.
URL: https://nda.nih.gov/